CLINICAL TRIAL: NCT02435355
Title: Efficiency of a Phone Coaching Program on Adherence to Continuous Positive Airway Pressure in Sleep Apnea Hypopnea Syndrome
Brief Title: Efficiency of a Phone Coaching for Sleep Apnea Hypopnea Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sadir Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Sadir Association
Record Dates: First submitted 2015-04-30; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep apnea; education; compliance; CPAP
MeSH Terms: conditions — Sleep Apnea Syndromes; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard support (No Intervention): All patients in this study underwent this procedure, which is the regular procedure in France.
- coached group (Experimental): In the coached group (CG), patients received standard support completed by 5 sessions (day 3, 10, 30, 60, 90 with equipment at home) of telephone-based counselling session by competent staff. Sessions were performed by a qualified person in education, qualifies by a university degree (Paul Sabatier University, Toulouse, France). The dates of phone calls were planned with the patient availabilities.
  Interventions: Behavioral: telephone-based counselling

INTERVENTIONS:
Behavioral: telephone-based counselling — The objective of the first session was to assess the patient's knowledge about the disease, device and health consequences. The importance of good adherence was emphasized, encouraging the patients to use the CPAP device throughout sleep every day. Objectives of the other educational sessions were first to identify disadvantages or obstacles to follow CPAP treatment and then focus on the benefits linked to use of CPAP. A particular effort was made to discuss misconceptions about sleep apnea and barriers to use, concerns fears and beliefs, as well as the perceptions of their partners and family, in order to increase patients' positive expectations regarding CPAP benefits.
  Arms: coached group

SUMMARY:
Background: Continuous Positive Airway Pressure (CPAP) remains the reference treatment for moderate to severe forms of the Sleep Apnea/Hypopnea Syndrome (SAHS). Compliance to the treatment appears to be a key factor to improving health status of these patients.

Methods: The investigators conducted a multicenter, prospective, randomized, controlled, parallel group trial of standard support completed or not within 3 months of coaching sessions for newly diagnosed SAHS patients starting CPAP therapy. The coaching session consisted of 5 sessions of telephone-based counseling by competent staff. The primary outcome was the proportion of patients using CPAP more than 3 hours per night for 4 months; the secondary outcome was mean hours of CPAP usage in the 2 groups.

DETAILED DESCRIPTION:
We conducted a multicenter, prospective, randomized, controlled, parallel group trial of standard support versus phone coaching for newly diagnosed SAHS patients starting CPAP therapy. Patients for clinical polysomnographic evaluation were recruited from April 2010 to March 2012. Those who were subsequently diagnosed with SAHS and prescribed CPAP were included in the study. The patient population was then randomized into two groups, one that received standard CPAP support only and the other standard support completed by a coaching session.

Procedure Standard support All patients in this study underwent this procedure, which is the regular procedure in France. In short, the patient received information by their physician, about modalities and usefulness of CPAP treatment. In the week following this information, a technician from the home care provider (SADIR based in France) brought CPAP equipment to the home, re-explained the device function and checked the mask adaptation to the patient. The follow-up of the patient by the home care provider consisted of one visit at home the first month to check the mask's tolerance and the functioning of the machine. An other visit was performed after 4 months to assess CPAP parameters (length of use, mask leaks, and residual AHI). Sleep physician checked the compliance and efficiency of CPAP treatment once the first month, then at 3 and 6 months. The compliance was then assessed by patient questioning and by looking at the data registered by the machine. After this period, the medical follow up was performed once a year.

Coached group In the coached group (CG), patients received standard support completed by 5 sessions (day 3, 10, 30, 60, 90 with equipment at home) of telephone-based counselling session by competent staff. Sessions were performed by a qualified person in education, qualifies by a university degree (Paul Sabatier University, Toulouse, France). The dates of phone calls were planned with the patient availabilities.

The objective of the first session was to assess the patient's knowledge about the disease, device and health consequences. The importance of good adherence was emphasized, encouraging the patients to use the CPAP device throughout sleep every day. Objectives of the other educational sessions were first to identify disadvantages or obstacles to follow CPAP treatment and then focus on the benefits linked to use of CPAP. A particular effort was made to discuss misconceptions about sleep apnea and barriers to use, concerns fears and beliefs, as well as the perceptions of their partners and family, in order to increase patients' positive expectations regarding CPAP benefits. The qualified person in education could also refer any problems in links with SAHS encountered by the patient to the technician, psychologist or dietician (employed by the home care provider). They can respectively help the patient with CPAP technical advice, mentally blocked with CPAP or diet counseling. The average length of each phone call was approximately 15 to 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed with SAHS
* CPAP treatment prescribed

Exclusion Criteria:

* previously use CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
proportion of patients using Continuous Positive Airway Pressure for more than 3 hours per night in the 2 groups | CPAP use was evaluated for 4 months

REFERENCES:
- [Derived] Sedkaoui K, Leseux L, Pontier S, Rossin N, Leophonte P, Fraysse JL, Didier A. Efficiency of a phone coaching program on adherence to continuous positive airway pressure in sleep apnea hypopnea syndrome: a randomized trial. BMC Pulm Med. 2015 Sep 14;15:102. doi: 10.1186/s12890-015-0099-7. PMID 26370444